CLINICAL TRIAL: NCT03892681
Title: Hepatocyte-specific Versus Extracellular Contrast Agents for Liver MRI: Prospective, Intra-individual Comparison of Diagnostic Performance for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2018-1047
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis; Liver Cirrhosis
Keywords: HBsAg(+) with chronic hepatitis or cirrhosis; anti-HCV(+) with cirrhosis; cirrhosis of any etiology
MeSH Terms: conditions — Hepatitis, Chronic; Liver Cirrhosis; Hepatitis B; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- contrast agents for liver MRI (Other)
  Interventions: Other: hepatocyte-specific contrast agent, extracellular contrast agent

INTERVENTIONS:
Other: hepatocyte-specific contrast agent, extracellular contrast agent — The type of contrast agent for the 1st MRI will be performed using hepatocyte-specific contrast agent (Primovist). The participant will undergo the 2nd MRI using extracellular contrast agent (Gadovist).

SUMMARY:
Adult patients with chronic hepatitis B and cirrhosis of any etiology who are found to have suspected liver cancer are potentially eligible for the study. All enrolled patients will undergo two MRI scans using two different contrast agents. The type of contrast agent for the 1st MRI will be performed using hepatocyte-specific contrast agent. The participant will undergo the 2nd MRI using extracellular contrast agent. The MRI examinations will be independently interpreted by two different radiologists. The radiologists will evaluate focal hepatic lesions and categorize them according to the LI-RADS v2018 and EASL 2018. Once the diagnosis is made, the participants will be provided with the standard of care. After the initial treatment, the participants will be followed up with multi-phasic dynamic contrast-enhanced CT every 3 or 6 months for at least 2 years. Based on the prospectively written radiology reports, the diagnostic performances will be calculated and compared between MRI with hepatocyte-specific contrast agent and MRI with extracellular contrast agent, using the pathology and clinical criteria as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 20 years
2. HBsAg (+) with chronic hepatitis or cirrhosis, anti-HCV (+) with cirrhosis, or cirrhosis of any etiology

   * The presence of cirrhosis will be determined based on the histologic or radiologic findings, including liver surface nodularity, margin blunting, segmental hypertrophy/atrophy, and findings secondary to portal hypertension (i.e., splenomegaly, esophageal or gastric varices, ascites, or reverse portal vein flow).
3. Child-Pugh class A or B
4. Up to three suspicious focal lesions between 10 mm and 30 mm found on US, CT, or MRI

   * Patients with a history of HCC treated by surgery or tumor ablation could be included, but only new nodules at a distance of > 2 cm from previously treated lesions were considered.

Exclusion Criteria:

1. Currently pregnant or lactating
2. Risk group for the use of gadolinium-enhanced MRI including severely decreased renal function (stage 4 or 5 chronic renal failure with eGFR ˂ 30 mL/min/1.73 m2), claustrophobia
3. Patients with history of chemoembolization or systemic treatment for liver cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | an expected average of 2 weeks
  The comparison of sensitivity between MRI using hepatocyte-specific contrast agent and extracellular contrast agent in the diagnosis of hepatocellular carcinoma The per-lesion sensitivity will be compared using McNemar's test.
Specificity | an expected average of 2 weeks
  The comparison of specificity between MRI using hepatocyte-specific contrast agent and extracellular contrast agent in the diagnosis of hepatocellular carcinoma.
  The per-lesion sensitivity will be compared using McNemar's test.

SECONDARY OUTCOMES:
Inter-reader agreement between two radiologists | an expected average of 2 weeks
  The inter-reader agreement between two radiologists for the LI-RADS v2018 categorization and diagnosis of HCC according to EASL 2018 in each MRI using hepatocyte-specific contrast agent and extracellular contrast agent.
  The inter-reader agreement will be evaluated using Cohen κ coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No